CLINICAL TRIAL: NCT05461573
Title: A Phase 3, Multi-Center, Non-Comparative Study to Evaluate the Contraceptive Efficacy, Safety, and Tolerability of LPRI-CF113 Administered Orally for 13 Medication Cycles
Brief Title: Efficacy, Safety, and Tolerability of LPRI-CF113 as an Oral Contraceptive in Females
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insud Pharma (Industry)
Collaborators: Chemo Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CF113-303
Record Dates: First submitted 2022-06-30; First posted 2022-07-18 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Contraception; Change in Bone Mineral Density
Keywords: Contraceptive Method Switching
MeSH Terms: conditions — Contraception Behavior | interventions — drospirenone

STUDY DESIGN:
Intervention Model Description: All subjects enrolled in the study will participate in Part A of the study and receive the experimental drug LPRI-CF113 (drospirenone). Part A will investigate the efficacy, safety, and tolerability of LPRI-CF113.
  A subgroup of subjects that are age 18-45 and without further exclusion criteria to Part B will be enrolled in Part B of the study. Part B of the study will investigate the effects of LPRI-CF113 on bone mineral density.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A - An investigation of the efficacy, safety, and tolerability of LPRI-CF113 (Experimental): All subjects enrolled in the study will participate in Part A of the study. Part A of the study will investigate the efficacy, safety, and tolerability of LPRI-CF113.
  Interventions: Drug: Drospirenone
- Part B - The effect of LPRI-CF113 on bone mineral density in a subgroup age 18-45 (Experimental): A subgroup of subjects from Part A that are age 18-45 and without further exclusion criteria to Part B will be enrolled in Part B of the study. Part B of the study will investigate the effects of LPRI-CF113 on bone mineral density.
  Interventions: Drug: Drospirenone

INTERVENTIONS:
Drug: Drospirenone — LPRI-CF113 consists of 24 active white tablets containing drospirenone (DRSP) 4 mg followed by 4 active pink tablets containing DRSP 2.8 mg, taken orally once daily for 28 consecutive days, in consecutive cycles for 12 months (13 medication cycles) without a break in daily tablet intake.
  Other Names: LPRI-CF113

SUMMARY:
This study will be in two parts, Part A and Part B. The primary objective of Part A is to evaluate the contraceptive efficacy of LPRI-CF113. The secondary objective of Part A is to evaluate the safety and tolerability of LPRI-CF113. The primary objective of Part B is to evaluate the impact of LPRI-CF113 on bone mineral density (BMD) at the lumbar spine (L1-L4) after 12 months (13 medication cycles). The secondary objective of Part B is to evaluate the impact of LPRI-CF113 on BMD and bone turnover after 12 months (13 medication cycles) at the femoral neck, total hip, and total body.

DETAILED DESCRIPTION:
This is a Phase 3, prospective, multi-center, open-label, non-comparative study in female subjects 13 to 45 years of age (inclusive) to determine the efficacy, safety, and tolerability of LPRI-CF113 administered orally for 13 (28-day) medication cycles (Part A). Healthy, sexually active female subjects of childbearing potential, who present to the clinic seeking contraception, will be enrolled in the study.

Part B will be an investigation of bone mineral density (BMD) at the lumbar spine and BMD and bone turnover at the femoral neck, total hip, and total body. Part B will consist of a subgroup of subjects enrolled in Part A (i.e., subjects that meet all of Part A inclusion criteria and none of Part A AND Part B exclusion criteria) who are 18 to 45 years of age (inclusive at the time of screening). BMD will be assessed by dual-energy X-ray absorptiometry (DXA) scan.

The study duration (Parts A and B) for each subject will be up to approximately 404 days (28 days [screening] + 376 days [Treatment and Follow-up Period]), unless the subject meets criteria for the extended Part B Follow-up, in which the duration will be approximately 769 days (28 days [screening] + 376 days [Treatment and Follow-up Period] + 365 days [extended Part B Follow up]).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to provide written informed consent (for adults) or assent (for adolescents <18 years of age) and comply with all study procedures, prohibitions, restrictions, and scheduled visits
* Subjects must be female, healthy, sexually active, postmenarcheal, premenopausal, and of childbearing potential, between 13 and 45 years of age (inclusive at the time of screening) and at risk for pregnancy

  * Note: Childbearing potential is defined as subjects who are ovulating, premenopausal, and not surgically sterile (ie, have not undergone hysterectomy, salpingectomy, or bilateral oophorectomy). Subjects that have undergone unilateral oophorectomy will not be considered surgically sterile and may be included in the study
  * Note: Only subjects 18 to 45 years of age (inclusive at the time of screening) are eligible for inclusion in Part B
* Subjects must be willing to have vaginal intercourse (with a genetically male partner) throughout the Treatment Period (ie, during each medication cycle) without using a secondary (eg, spermicides) or emergency method of contraception
* Subjects must have a BMI of 18 kg/m2 or higher
* Subjects must have a systolic blood pressure of 159 mmHg or lower and a diastolic blood pressure of 99 mmHg or lower

  * Note: The median of 3 blood pressure measurements will be used for this criterion
  * Note: Subjects are required to rest for 5 minutes prior to the first blood pressure measurement and for 1 minute between subsequent measurements. Measurements done without appropriate preparation of the subject (excluding caffeine use, smoking, or excessive physical activity) should not be considered, and the measurement should be repeated upon appropriate preparation of the subject
* Subjects must be regularly menstruating (with cycle length between 21 and 35 days) for at least 3 months prior to the signing of the Informed Consent Form

  * Note: Breastfeeding women can be included 6 weeks after delivery irrespective of menstrual cycles post-delivery
* Subjects must agree to not use any secondary (eg, spermicides) or emergency contraceptive methods during the study period
* Subjects must not be enrolled or plan to enroll in any other clinical study during the study period
* Subjects must be willing to use the study drug (LPRI-CF113) for 13 (28-day) medication cycles, and be willing to use the provided diary
* Subjects must generally be in good physical and mental health based on a medical history and a physical examination performed by the Investigator at screening

Exclusion Criteria:

PART A:

* The subject is pregnant at the time of screening
* The subject has a desire to become pregnant at the time of screening

  * Note: The subject will be asked if she has a desire for pregnancy at screening (and at each study visit). If a positive answer is given at screening, the subject will be excluded
* The subject plans regular concomitant use of barrier contraceptive methods, spermicides, intrauterine device, other contraceptive measures, prohibited medications, and drugs contraindicated for study drug
* The subject has an abnormal and clinically significant finding on pelvic, breast, or ultrasound examination at screening based on the judgment of the Investigator
* The subject has an abnormal and clinically significant finding on physical examination, clinical laboratory assessments (chemistry, hematology, urinalysis), or 12-lead ECG assessment based on the judgment of the Investigator
* The subject has had less than 3 menstrual cycles after discontinuing dosing of depot medroxyprogesterone acetate (Depo-Provera®) or any combined injectable contraceptive (eg, Cyclofem®) prior to consent/assent. Those with spontaneous menses while on injectable contraceptive will be considered for inclusion
* The subject has received any of the following:

  * A progestin-releasing intra-uterine device or contraceptive implant within 2 months prior to screening or
  * A beta-human chorionic gonadotropin (β-hCG) or co-medication containing β-hCG within 1 month prior to screening
* The subject at the time of screening has a history of primary amenorrhea or secondary amenorrhea (with or without known etiology)

  * Note: Primary amenorrhea is defined as no menarche by 16 years of age with normal secondary sexual characteristics
  * Note: Secondary amenorrhea is defined as the absence of menses for 3 months in the setting of previously normal (ie, regular) menstruation
* The subject has a current male sexual partner with a history of infertility, vasectomy, or bilateral orchiectomy
* The subject has an abnormal Pap smear finding of low-grade squamous intraepithelial lesion or higher at screening or 6 months prior to screening. Subjects <21 years of age at screening do not require a Pap smear

  * Note: Human papilloma virus (HPV) testing, by polymerase chain reaction (PCR), will be performed only in the case of atypical squamous cells of undetermined significance (ASC-US). Subjects with ASC-US can be included if negative for high-risk HPV strains
  * Note: A historical Pap smear may be used for eligibility if performed within the past 6 months with results available
* The subject has a history of uncontrolled medical illness (eg, the subject has an uncontrolled thyroid disorder and is not on a stable treatment regimen for 2 or more months)
* The subject has a history of jaundice while taking hormonal contraceptives
* The subject has a history of alcohol or substance use disorder within 12 months prior to screening. Alcohol abuse is defined as typical consumption of 14 or more alcoholic drinks weekly

  * Note: One drink of alcohol is equivalent to ½ pint of beer (285 mL), 1 glass of spirits (25 mL), or 1 glass of wine (125 mL)
* The subject has a history or current evidence of clinically significant psychiatric illness, such as major depression or schizophrenia, that in the opinion of the Investigator contraindicates participation in the study
* The subject has surgical procedures scheduled to occur during the study that would preclude use of contraceptives or require withdrawal of contraceptives
* The subject has a history of an inherited or acquired disorder that predisposes the subject to venous or arterial thromboembolism (eg, factor V Leiden mutation, prothrombin mutation, presence of antiphospholipid antibodies)
* The subject has received an investigational product within 3 months prior to screening
* The subject has a history of using or currently uses any medications known to interfere with the efficacy of hormonal contraceptives, or other prohibited medications or products
* Medications known to reduce the efficacy of hormonal contraceptives:

  * Barbiturates
  * Bosentan
  * Anticonvulsants (e.g., topiramate, phenytoin, carbamazepine, oxcarbazepine, felbamate, rufinamide)
  * Primidone
  * Rifampin
  * Human immunodeficiency virus peptidase inhibitors (e.g., ritonavir, nelfinavir)
  * Non-nucleoside reverse transcriptase inhibitors (e.g., nevirapine, efavirenz)
  * Griseofulvin
  * Products containing St. John's Wort (hypericum perforatum)
* Other prohibited medications or products:

  * Rifabutin
  * Aprepitant
  * Hepatitis C treatments (eg, boceprevir, telaprevir)
  * Azole antifungals (eg, fluconazole, itraconazole, ketoconazole, voriconazole)
  * Macrolides (eg, clarithromycin, erythromycin)
  * Verapamil
  * Diltiazem
  * Cyclosporine
  * Lamotrigine
  * Sex hormones
  * Grapefruit juice
* The subject has a history of severe or critical Coronavirus Disease 2019 (COVID-19) or has been hospitalized for COVID-19 within 3 months prior to screening

  * Note: Severe COVID-19 severity is defined as individuals who have SpO2 <94% on room air at sea level, a PaO2/FiO2 <300 mmHg, a respiratory rate >30 breaths/min, or lung infiltrates >50%
  * Note: Critical COVID-19 severity is defined as individuals who have respiratory failure, septic shock, and/or multiple organ dysfunction
* The subject has any ongoing condition or history of medical illness that in the opinion of the Investigator may jeopardize the conduct of the study or impact screening
* The subject is employed by the Sponsor, the Contract Research Organization (CRO), or the clinical facility (permanent, temporary contract worker, or designee responsible for the conduct of the study), or is a family member (spouse, parent, sibling, or child) of the Sponsor, CRO, or clinical facility employee
* The subject has a known contraindication or hypersensitivity to ingredients or excipients of the study drug (LPRI-CF113)
* The subject has a history of or is currently being treated for any of the following:

  * Renal insufficiency
  * Hepatic insufficiency
  * Adrenal insufficiency
  * Venous thromboembolism (ie, deep vein thrombosis, pulmonary embolism)
  * Arterial thromboembolism of cardiac origin (eg, valvular heart disease)
  * Cerebral vascular disease
  * Coronary artery disease
  * Diabetic vasculopathy
  * Headaches with focal neurological symptoms
  * Major surgery requiring more than 7 days of immobilization within 3 months prior to screening
  * Carcinoma of the breast
  * Estrogen or progestin sensitive malignancies
  * Abnormal vaginal bleeding in the 6 months prior to screening
  * Cholestatic jaundice during pregnancy
  * Liver tumor (benign or malignant)
  * Active liver disease
  * Rheumatoid arthritis

PART B:

* The subject is <18 years of age, inclusive
* The subject has a BMD Z-score of -1.5 at or lower at screening
* The subject has a history of low-trauma fracture (eg, fracture from a fall from standing height). This does not include fractures of the fingers, toes, or skull
* The subject has a history of medical conditions or procedures associated with low BMD. This includes the following:

  * Metabolic bone disease (eg, Paget's Disease of the bone, osteomalacia)
  * Collagen vascular disease (eg, Marfan syndrome, Ehlers-Danlos syndrome, osteogenesis imperfecta)
  * Malabsorptive disease (eg, inflammatory bowel disease, postgastrectomy syndrome)
  * Bariatric surgery (except gastric banding)
  * Abnormal bone mineral metabolism (eg, hypocalcemia/hypercalcemia, hypophosphatemia/hyperphosphatemia, hypomagnesemia)
* The subject has a history of chronic (3 or more months) use within 12 months of screening of the following medications known to increase BMD:

  * Bisphosphonates
  * Denosumab
  * Teriparatide
  * Abaloparatide
  * Romosozumab
  * Calcitonin
  * Fluoride
  * Strontium
* The subject has a history of chronic (3 or more months) use within 12 months of screening of the following medications known to decrease BMD:

  * Glucocorticoids administered orally, intravenously, or by inhalation.
  * Note: Subjects taking chronic oral or intravenous glucocorticoids (eg, prednisone >2.5 mg daily for 3 or more months) will have a washout period of 12 months
  * Depo-Provera.
  * Note: Subjects using Depo-Provera for 2 or more years will be excluded
  * Aromatase inhibitors within 2 years prior to screening
  * Raloxifene within 2 years prior to screening
  * Anticonvulsants (phenytoin, phenobarbital, carbamazepine, or valproate)
  * Protease inhibitors
  * Cyclosporine
  * Heparin
  * Warfarin
  * Thiazolidinediones
  * Sodium-glucose transporter protein 2 inhibitors
  * Tricyclic antidepressants
  * Proton pump inhibitors
  * Selective serotonin reuptake inhibitors within 3 months prior to screening
* The subject has any of the following that may preclude accurate BMD measurement by DXA scan:

  * History of lumbar spine surgery
  * History of bilateral hip surgery
  * Surgical placement of metallic implant (eg, nails, clips, screws, rods, pins, wires)
  * Piercings that cannot be removed
  * Weight or height that exceeds the limit of DXA scan table

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1542 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Part A (Efficacy Assessment): Number of pregnancies in subjects ≤35 years of age (at the time of screening). | 12 months
  Calculated by Pearl Index.

SECONDARY OUTCOMES:
Part A (Efficacy Assessment): Number of pregnancies from exposure cycles in subjects ≤35 years of age. | 12 months
  Calculated by Pearl Index.
Part A (Efficacy Assessment): Number of pregnancies from method failures in subjects ≤35 years of age. | 12 months
  Calculated by Pearl Index.
Part A (Efficacy Assessment): Pregnancy ratio from evaluable cycles, exposure cycles, and perfect cycles in subjects ≤35 years of age. | 12 months
  Calculated by life table analysis.
Part A (Efficacy Assessment): Number of pregnancies from exposure cycles, method failures, and evaluable cycles in all subjects. | 12 months
  Calculated by Pearl Index.
Part A (Efficacy Assessment): Pregnancy ratio in all subjects. | 12 months
  Calculated by life table analysis.
Part A (Efficacy Assessment): Number of pregnancies from exposure cycles, method failures, and evaluable cycles in subjects >35 years of age. | 12 months
  Calculated by Pearl Index.
Part A (Efficacy Assessment): Pregnancy ratio in subjects >35 years of age. | 12 months
  Calculated by life table analysis.

OTHER OUTCOMES:
Part A (Primary Safety Assessment): Incidence and severity of adverse events (AEs), adverse events of special interest (AESIs), drug-related AEs, and treatment-emergent AEs. | 12 months
  Can be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of the intervention drug (LPRI-CF113). Counts and percentages of subjects with AEs will be presented by system organ class and preferred term with the severity reported.
Part A (Primary Safety Assessment): Incidence and severity of abnormal clinical findings on physical examination, gynecological examination, and transvaginal ultrasound examination. | 12 months
  The investigator will exercise his or her clinical judgement in deciding whether an abnormal assessment is clinically significant. The incidence and severity of abnormal clinical findings will be summarized with counts and percentages.
Part A (Primary Safety Assessment): Incidence and severity of mastodynia/mastalgia and dysmenorrhea. | 12 months
  The incidence and severity of abnormal clinical findings will be summarized with counts and percentages.
Part A (Primary Safety Assessment): Incidence and severity of abnormal cervical cytology. | 12 months
  Assessed by pap smear.
Part A (Primary Safety Assessment): Incidence and severity of abnormal bleeding. | 12 months
  The number of bleeding or spotting days will be summarized by medication cycle. The number of bleeding or spotting episodes, length of bleeding or spotting episodes, number of subjects with prolonged bleeding (>14 days in a 90-day reference period), and incidence of unscheduled bleeding will be summarized.
Part A (Primary Safety Assessment): Incidence of clinical laboratory abnormalities from baseline, including chemistry, hematology, and urinalysis, considered significant by the Investigator. | 12 months
  Incidence of laboratory abnormalities will be summarized with counts and percentages.
Part A (Primary Safety Assessment): Incidence of vital sign abnormalities from baseline, including blood pressure, heart rate, respiratory rate, and body temperature, considered significant by the Investigator. | 12 months
  Absolute values and changes from baseline of vital signs will be summarized using descriptive statistics.
Part A (Primary Tolerability Assessment): Changes in quality of life. | 12 months
  Assessed by Q-LES-Q-SF (Quality of Life, Enjoyment, and Satisfaction Questionnaire-Short Form)
Part A (Primary Tolerability Assessment): Acceptability of study drug. | 12 months
  All subjects will be asked by the Investigator via questionnaire: Are you satisfied with this oral contraceptive method? For subjects who suspended their oral contraceptive method in order to begin administration of the study drug, the Investigator will ask: How was your wellbeing during the intake of the study drug in comparison to the time when you took your formal contraceptive?
Part B (Primary Safety Assessment): Mean percentage change in lumbar spine (L1-L4) bone mineral density (BMD) in subjects ≥18 years of age. | Baseline to 12 months
  BMD measured by dual-energy X-ray absorptiometry (DXA) scan.
Part B (Secondary Safety Assessment): Mean absolute changes in lumbar spine (L1-L4) BMD in subjects ≥18 years of age. | Baseline to 12 months
  BMD measured by DXA scan.
Part B (Secondary Safety Assessment): Mean absolute and percentage changes in BMD (femoral neck, total hip, and total body) in subjects ≥18 years of age. | Baseline to 12 months
  BMD measured by DXA scan.
Part B (Secondary Safety Assessment): Mean absolute and percentage changes in BMD (lumbar spine, femoral neck, total hip, and total body) in subjects ≥18 years of age. | Baseline to 6 months
  BMD measured by DXA scan.
Part B (Secondary Safety Assessment): Mean absolute changes in BMD Z-scores (lumbar spine, femoral neck, total hip, and total body) in subjects ≥18 years of age. | Baseline to 6 months and 12 months
  BMD measured by DXA scan.
Part B (Secondary Safety Assessment): Proportion of subjects with percentage changes in lumbar spine, femoral neck, total hip, and total body BMD by categories in subjects ≥18 years of age. | Baseline to 12 months
  BMD measured by DXA scan, categories defined as ≥0%, <0% to -1.5%, <-1.5% to -3%, <-3% to -5%, <-5% to -8%, and <-8%.
Part B (Secondary Safety Assessment): Proportion of subjects with absolute changes in BMD Z-scores (lumbar spine, femoral neck, total hip, and total body) in subjects ≥18 years of age. | Baseline to 6 months and 12 months
  BMD measured by DXA scan, categories defined as ≥0.5, <0.5 to 0.3, <0.3 to 0, <0 to -0.3, <-.3 to -0.5, and <-0.5.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Colli, MD, Study Director — Chemo Research SL
Locations (47):
- United States (46):
  - Alabama Clinical Therapeutics, LLC, Alabaster, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Del Sol Research Management, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Cornerstone Research Institute - Longwood, Altamonte Springs, Florida
  - Encore Medical Research of Boynton Beach LLC., Boynton Beach, Florida
  - Women's Medical Research Group, Clearwater, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Inpatient Research Clinic, LLC, Hialeah, Florida
  - Vital Pharma Research, Inc., Hialeah, Florida
  - Encore Medical Research, LLC, Hollywood, Florida
  - Global Research Associates, Homestead, Florida
  - Altus Research, Lake Worth, Florida
  - Florida International Medical Research, Miami, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - SJ Research Institute, Miami, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - American Research Centers of Florida, Pembroke Pines, Florida
  - Comprehensive Clinical Trials, West Palm Beach, Florida
  - Encore Medical Research of Weston LLC, Weston, Florida
  - Fellows Research Alliance, Savannah, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - Rosemark WomenCare Specialists, Idaho Falls, Idaho
  - Praetorian Pharmaceutical Research, Marrero, Louisiana
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Eastern Clinical Research Associates, New Orleans, Louisiana
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Unified Women's Clinical Research - Raleigh, Raleigh, North Carolina
  - Unified Women's Clinical Research - Winston-Salem, Winston-Salem, North Carolina
  - Clinohio Research Services, Columbus, Ohio
  - AC Clinical Research, Tiffin, Ohio
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - The Research Center of the Upstate, Greenville, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - Discovery Clinical Trials, Dallas, Texas
  - TMC Life Research, Houston, Texas
  - FMC Science, Lampasas, Texas
  - Maximos OB/GYN, League City, Texas
  - Austin Regional Clinic ARC Clinical Research at Kelly Lan, Pflugerville, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Mt. Olympus Medical Research- Sugar Land Texas, Sugar Land, Texas
  - Eastern Virginia Medical School (EVMS), Norfolk, Virginia
  - Virginia Women's Health Associates, Reston, Virginia
- Clinique RS, Québec, Canada

REFERENCES:
- [Background] Rosenbaum P, Schmidt W, Helmerhorst FM, Wuttke W, Rossmanith W, Freundl F, Thomas K, Grillo M, Wolf A, Heithecker R. Inhibition of ovulation by a novel progestogen (drospirenone) alone or in combination with ethinylestradiol. Eur J Contracept Reprod Health Care. 2000 Mar;5(1):16-24. doi: 10.1080/13625180008500376. PMID 10836659
- [Background] SLYND (drospirenone) [prescribing information]. Florham Park, NJ. Exeltis USA, Inc. May 2019.
- [Background] Investigator's Brochure for Drospirenone Only Pill - LF111. Edition No. 12.0, 18 March 2021.
- [Background] Cibula D, Skrenkova J, Hill M, Stepan JJ. Low-dose estrogen combined oral contraceptives may negatively influence physiological bone mineral density acquisition during adolescence. Eur J Endocrinol. 2012 Jun;166(6):1003-11. doi: 10.1530/EJE-11-1047. Epub 2012 Mar 21. PMID 22436400
- [Background] Beksinska ME, Smit JA. Hormonal contraception and bone mineral density. Expert Rev of Obstet Gynecol. 2011;6(3):305-319.
- [Background] Investigator's Brochure for Drospirenone 4 mg and 2.8 mg Oral Tablets - LPRI-CF113. Edition No. 2.2, 10 August 2022.
- [Background] Thomas SL, Ellertson C. Nuisance or natural and healthy: should monthly menstruation be optional for women? Lancet. 2000 Mar 11;355(9207):922-4. doi: 10.1016/S0140-6736(99)11159-0. No abstract available. PMID 10752720
- [Background] Burkman R, Bell C, Serfaty D. The evolution of combined oral contraception: improving the risk-to-benefit ratio. Contraception. 2011 Jul;84(1):19-34. doi: 10.1016/j.contraception.2010.11.004. Epub 2010 Dec 24. PMID 21664507
- [Background] Bitzer J. Hormone withdrawal-associated symptoms: overlooked and under-explored. Gynecol Endocrinol. 2013 Jun;29(6):530-5. doi: 10.3109/09513590.2012.760194. Epub 2013 Feb 20. PMID 23421366
- [Background] Belsey EM, Machin D, d'Arcangues C. The analysis of vaginal bleeding patterns induced by fertility regulating methods. World Health Organization Special Programme of Research, Development and Research Training in Human Reproduction. Contraception. 1986 Sep;34(3):253-60. doi: 10.1016/0010-7824(86)90006-5. PMID 3539509